CLINICAL TRIAL: NCT05254756
Title: "A Comparison of the Bouquet Speculum and the Traditional 2-Bladed Speculum"
Brief Title: "Pilot Study: A Comparison of the Bouquet Speculum and the Traditional 2-Bladed Speculum"
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because of logistical issues with the sites.
Sponsor: Isain Zapata (Other)
Responsible Party: Sponsor-Investigator, Isain Zapata, Assistant Professor in Research and Statistics, Rocky Vista University, LLC
Organization: Rocky Vista University, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB #2020--0110
Record Dates: First submitted 2022-02-04; First posted 2022-02-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pelvic Exam

STUDY DESIGN:
Intervention Model Description: This randomized single-blinded clinical study
Who Masked: Participant, Care Provider
Masking Description: Patients who have an indication for a speculum exam and who meet other inclusion criteria will be randomized to either receive their exam with the traditional plastic 2-blade disposable speculum or the 5-petal Bouquet speculum. After the exam, the patient and the physician will each fill out a questionnaire that will ask about patient comfort, ease of use, visibility of the cervix, and perceived time of the exam.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional plastic 2-blade disposable speculum (Active Comparator): Patients assigned to this arm will be evaluated using the traditional plastic 2-blade disposable speculum
  Interventions: Device: Traditional plastic 2-blade disposable speculum
- 5-petal Bouquet speculum (Experimental): Patients assigned to this arm will be evaluated using the 5-petal Bouquet speculum
  Interventions: Device: Bouquet speculum

INTERVENTIONS:
Device: Bouquet speculum — Quantitative assessments of visualization of cervix, ease-of-use by the provider, and comfort of the patient
  Other Names: 884.4520
  Arms: 5-petal Bouquet speculum
Device: Traditional plastic 2-blade disposable speculum — Quantitative assessments of visualization of cervix, ease-of-use by the provider, and comfort of the patient
  Arms: Traditional plastic 2-blade disposable speculum

SUMMARY:
This randomized single-blinded clinical study will compare the typical 2-bladed plastic disposable vaginal speculum to the novel 5-petal Bouquet speculum on level of patient comfort, visibility of the cervix, and time length of the examination. The data will be collected via patient and provider questionnaires.

DETAILED DESCRIPTION:
For nearly 200 years, the traditional 2-blade "Duck bill" vaginal speculum has had very little evolution in design. In past decades, there has been an increase in popularity in using the plastic speculum rather than the metal speculum. The plastic speculum has effectively the same design as the traditional metal vaginal speculum. The current 2-blade design that has been used for centuries leaves many women feeling pain or discomfort during a speculum vaginal exam. Furthermore, in obese and multiparous women, the 2-blade design often allows the lateral walls of the vagina to cave inward during the exam, preventing the provider from gaining full visibility of the cervix. Another common complaint is that the exam takes too long, which leaves patients in pain and feeling vulnerable for an extended period of time.

The novel 5-petal Bouquet vaginal speculum offers an alternative design that some have argued provides enhanced patient comfort, better visualization of the cervix, and is easier to use for the provider. This proposed study design is a blueprint that will be used to compare the Bouquet speculum to a traditional 2-blade disposable plastic speculum on patient comfort, visualization of the cervix, and ease of use for the provider. The investigators predict that the results of this study will help physicians and other medical providers provide patients with better experience, reducing or eliminating the current common complaints regarding how speculum exams are performed today.

ELIGIBILITY:
Inclusion Criteria:

* Female patients that require a pelvic exam.
* 18 years of age or older
* Having had at least one previous pelvic exam with the traditional speculum
* Consent to participate in the study

Exclusion Criteria:

- Never had a pelvic exam before

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Patient comfort | Immediately after the exam
  Find the difference in the level of patient comfort during a vaginal speculum exam between the traditional 2-blade plastic disposable speculum and the 5-petal Bouquet speculum.
  Assessed with a questionnaire answered by the patient:
  1. What was the level of comfort with this Pap smear compared to other speculum exams you have had? (More comfortable, Same level of comfort/discomfort, Less comfortable )
  2. Based on what you anticipated the exam was:
     (More comfortable, As comfortable/uncomfortable, Less comfortable)
  3. On a scale from 0 to 10, what is the highest level of pain you experienced during the Pap smear/speculum exam? (10 being the worst pain you have ever experienced, and 0 being no pain)
  4. Did the doctor who performed the exam ask you adjust your body position while the speculum was inserted? (Yes, No)
  5. What is your estimation of how long the speculum was inserted? (0-30 seconds, 30-60 seconds, 1-2 minutes, 2-3 minutes, >3 minutes)
Length of time | During the exam
  Find the difference in the length of time that the Bouquet speculum is inserted during a Pap smear compared to the traditional 2-blade speculum.
  The time the speculum is inserted is recorded for every interactions.
Ease of use | Immediately after the exam
  Find the difference in ease of use for the provider between the traditional 2-blade plastic disposable speculum and the 5-petal Bouquet speculum.
  Assessed with a questionnaire answered by the provider:
  1. During the speculum exam, were the lateral walls of the cervix easily visualized upon initial visualization of the cervix? (Yes, No)
  2. What is your estimate of how long the speculum was inserted? (0-30 seconds, 30-60 seconds, 1-2 minutes, 2-3 minutes, >3 minutes)
  3. While the speculum was inserted, was the patient asked to adjust body position in order to gain a better view of the cervix? (Yes, No)
  4. Were special maneuvers performed in order to better visualize the cervix? (e.g. use a different size/type of speculum, apply a condom over the speculum to view the lateral walls, re-insert the speculum, etc.)? (Yes, No)

CONTACTS AND LOCATIONS:
Overall Officials: James M Small, MD, Principal Investigator — Rocky Vista University
Locations (1):
- St. George OB/GYN, St. George, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data will be shared when reasonable request is asked to the principal investigator. however this is yet to be decided.

REFERENCES:
- [Background] Bouquet JM, Chernau A, McLaughlin R, Choudhury Q. 2019. A New Vaginal Speculum and an Inexpensive Kit to Screen and Treat Dysplasia and Cancer of the Cervix. Journal of Women's Health Care. 8.470 doi: 10.35248/2167-0420.19.8.470